CLINICAL TRIAL: NCT02280265
Title: Evaluate Efficacy and Safety of ADVATE in the Standard Prophylaxis Treatment of Severe or Moderately Severe Hemophilia A.
Brief Title: Efficacy and Safety of ADVATE Standard Prophylaxis to Hemophilia A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yongjun Fang,MD, Director of Department of Hematology/Oncology, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prophylaxis201407008-1
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Hemophilia A
Keywords: hemophilia A; standard prophylaxis; Recombinant Human Coagulation Factor VIII for injection; ADVATE; Pediatric
MeSH Terms: conditions — Hemophilia A | interventions — Injections; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADVATE (Experimental): The baseline ABR will be assessed from bleeding log and clinic records from preceding year. Subjects will initially be treated standard prophylaxis(20 - 40 IU/Kg body weight every 48 ± 6 hours) with Recombinant Human Coagulation Factor VIII for injection(ADVATE) for 1 year. Subjects must be prescribed ADVATE by the treating physician. Data will be collected over a period of 2 years from the time of study enrollment. Study visits are to coincide with routinely rescheduled and emergency visits. Available data from these visits shall be transcribed onto the case report forms (CRFs).
  Interventions: Drug: Recombinant Human Coagulation Factor VIII for injection

INTERVENTIONS:
Drug: Recombinant Human Coagulation Factor VIII for injection — Subjects will initially be treated standard prophylaxis(20 - 40 IU/Kg body weight 2 times one week) with ADVATE for 1 year.
  Other Names: ADVATE

SUMMARY:
Hemophilia A is an X-linked recessive, congenital bleeding disorder caused by deficient or defective coagulation factor VIII (FVIII). Prophylaxis is recommended as the standard of care for boys with severe haemophilia by WHO and World Federation Of Hemophilia (WFH). The efficacy and safety of prophylaxis in preventing bleeds and arthropathy in patients with hemophilia has been confirmed in well-designed clinical studies.To keep the factor level above 1%, the standard dosage for patients with severe hemophilia A is 20-40 Units /kg/infusion (average 30 Units /kg) every other day or three times a week. This dosage has a very high consumption of factor, up to 5000-6000 international unit (IU)/kg/year. The high consumption of factor and cost present a major barrier to use the standard prophylaxis in many countries particularly in the developing world.

In China the majority of boys with severe hemophilia A can only pay for on-demand treatment or low-dose prophylaxis. Ao after the affordability of patients was solved and many patients will get more chance to receive standard prophylaxis.

This study is designed to evaluate the Annual Bleeding rate (ABR), joint health outcomes and QoL outcomes in subjects using ADVATE(Recombinant Human Coagulation Factor VIII for injection) standard prophylaxis under the conditions of routine practice.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has hemophilia A with FVIII≤2 %.
2. Previously treated patients (PTPs).
3. Age from 2 to 18 years.

Exclusion Criteria:

1. Subject has known hypersensitivity to the active substance or any of the excipients.
2. Subject has known allergic reaction to mouse or hamster proteins.
3. Subject has participated in another clinical study involving an investigational product (IP) or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving another FVIII concentrate or device during the course of this study.
4. Subject is planned, or likely to have surgery during the study period.
5. Subject has end-stage renal failure or evidence of a severe or uncontrolled systemic disease as judged by the investigator.
6. Subject has full-blown Acquired Immuno Deficiency Syndrome (AIDS),determined by Cluster Determinant 4+(CD4+) and clinical presentation.
7. Subject has active hepatic disease (alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels > 5 times the upper limit of normal).
8. Subject has clinical or laboratory evidence of severe liver impairment including (but not limited to) a recent and persistent international normalized ratio (INR)> 1.4, and/or the presence of splenomegaly and/or significant spider angioma on physical exam, and/or a history of esophageal hemorrhage or documented esophageal varices.
9. The subject in the opinion of the investigator is unable or unwilling to comply with study protocol
10. Subject is a family member of the investigator or site staff

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
ABR | 3 months
  To evaluate the Annual Bleeding rate (ABR) in subjects using standard prophylaxis under the conditions of routine practice.

SECONDARY OUTCOMES:
incidence of new target joints | 3 months
  Incidence of new target joints.
Pettersson score of joint | 3 months
  Status of joint health by X-ray using Pettersson score
magnetic resonance imaging scoring of joint | 6 months
  Status of joint health by magnetic resonance imaging scoring system.
Hemophilia Joint Health Score (HJHS) of joint | 3 months
  Status of joint health using HJHS
Number of ADAVTE units | 3 months
  Number of Recombinant Human Coagulation Factor VIII for injection (ADAVTE) units required for bleed cessation and Number of ADVATE infusions required for bleed cessation
QoL of patients wiht hemophilia | 3 months
  QoL assessment by Canadian Haemophilia Outcomes - Kids Life Assessment Tool (CHO-KLAT)
Inhibitor rate | 3 months
  Inhibitor rate monitoring: inhibitor will be tested at entry of study, every 3 months and at end of study.

REFERENCES:
- [Background] Astermark J, Petrini P, Tengborn L, Schulman S, Ljung R, Berntorp E. Primary prophylaxis in severe haemophilia should be started at an early age but can be individualized. Br J Haematol. 1999 Jun;105(4):1109-13. doi: 10.1046/j.1365-2141.1999.01463.x. PMID 10554828
- [Background] Berntorp E, Boulyjenkov V, Brettler D, Chandy M, Jones P, Lee C, Lusher J, Mannucci P, Peak I, Rickard K, et al. Modern treatment of haemophilia. Bull World Health Organ. 1995;73(5):691-701. PMID 8846496
- [Background] Manco-Johnson MJ, Abshire TC, Shapiro AD, Riske B, Hacker MR, Kilcoyne R, Ingram JD, Manco-Johnson ML, Funk S, Jacobson L, Valentino LA, Hoots WK, Buchanan GR, DiMichele D, Recht M, Brown D, Leissinger C, Bleak S, Cohen A, Mathew P, Matsunaga A, Medeiros D, Nugent D, Thomas GA, Thompson AA, McRedmond K, Soucie JM, Austin H, Evatt BL. Prophylaxis versus episodic treatment to prevent joint disease in boys with severe hemophilia. N Engl J Med. 2007 Aug 9;357(6):535-44. doi: 10.1056/NEJMoa067659. PMID 17687129
- [Background] Gringeri A, Lundin B, von Mackensen S, Mantovani L, Mannucci PM; ESPRIT Study Group. A randomized clinical trial of prophylaxis in children with hemophilia A (the ESPRIT Study). J Thromb Haemost. 2011 Apr;9(4):700-10. doi: 10.1111/j.1538-7836.2011.04214.x. PMID 21255253
- [Background] Valentino LA, Mamonov V, Hellmann A, Quon DV, Chybicka A, Schroth P, Patrone L, Wong WY; Prophylaxis Study Group. A randomized comparison of two prophylaxis regimens and a paired comparison of on-demand and prophylaxis treatments in hemophilia A management. J Thromb Haemost. 2012 Mar;10(3):359-67. doi: 10.1111/j.1538-7836.2011.04611.x. PMID 22212248
- [Background] Srivastava A, Brewer AK, Mauser-Bunschoten EP, Key NS, Kitchen S, Llinas A, Ludlam CA, Mahlangu JN, Mulder K, Poon MC, Street A; Treatment Guidelines Working Group on Behalf of The World Federation Of Hemophilia. Guidelines for the management of hemophilia. Haemophilia. 2013 Jan;19(1):e1-47. doi: 10.1111/j.1365-2516.2012.02909.x. Epub 2012 Jul 6. PMID 22776238
- [Background] Nilsson IM, Berntorp E, Lofqvist T, Pettersson H. Twenty-five years' experience of prophylactic treatment in severe haemophilia A and B. J Intern Med. 1992 Jul;232(1):25-32. doi: 10.1111/j.1365-2796.1992.tb00546.x. PMID 1640190
- [Background] Ljung R. Prophylactic therapy in haemophilia. Blood Rev. 2009 Nov;23(6):267-74. doi: 10.1016/j.blre.2009.08.001. Epub 2009 Sep 22. PMID 19775786